CLINICAL TRIAL: NCT03806413
Title: Post-surgical Delirium in Patients Undergoing Open Heart Surgery.
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohammad Hazem I. Ahmad Sabry, Lecturer of Anesthesia, University of Alexandria
Other Study IDs: 16/68(8/2/2017)
Record Dates: First submitted 2019-01-05; First posted 2019-01-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Delirium; Open Heart Surgery
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open heart surgery: The study will be done on patients undergoing open heart surgery in Alexandria University hospitals from January 5th 2019 till January 4th 2020. The 6-item Cognitive Impairment Test (6CIT) and SPMSQ questionnaire will be used. SPMSQ will be done preoperative and daily for 3 days postoperative, at day 7. Phone call for SPMSQ will be done 3, 6 9 and 12 months after surgery.
  Interventions: Other: Open heart surgery

INTERVENTIONS:
Other: Open heart surgery — The study will be done on patients undergoing open heart surgery in Alexandria University hospitals from January 5th 2019 till January 4th 2020. The 6-item Cognitive Impairment Test (6CIT) and SPMSQ questionnaire will be used. SPMSQ will be done preoperative and daily for 3 days postoperative, at day 7. Phone call for SPMSQ will be done 3, 6 9 and 12 months after surgery.
  Other Names: On-pump cardiac surgery

SUMMARY:
Post-surgical delirium in patients undergoing open heart surgery. Introduction Delirium occurs after open heart surgery may reach about 1/3 of the patients.(1)

Aim The aim of this study is to determine the incidence of delirium after open heart surgery and the associated risk factors in Alexandria University hospital.

Patients and Methods The study will be done on patients undergoing open heart surgery in Alexandria University hospitals from January 5th 2019 till January 4th 2020. The 6-item Cognitive Impairment Test (6CIT) and SPMSQ questionnaire will be used. SPMSQ will be done preoperative and daily for 3 days postoperative, at day 7. Phone call for SPMSQ will be done 3, 6 9 and 12 months after surgery.

DETAILED DESCRIPTION:
Post-surgical delirium in patients undergoing open heart surgery. Introduction Delirium occurs after open heart surgery may reach about 1/3 of the patients.(1)

Aim The aim of this study is to determine the incidence of delirium after open heart surgery and the associated risk factors in Alexandria University hospital.

Patients and Methods The study will be done on patients undergoing open heart surgery in Alexandria University hospitals from January 5th 2019 till January 4th 2020. The 6-item Cognitive Impairment Test (6CIT) and SPMSQ questionnaire will be used. SPMSQ will be done preoperative and daily for 3 days postoperative, at day 7. Phone call for SPMSQ will be done 3, 6 9 and 12 months after surgery.

Results Results will be collected in tables and graphs. Appropriate statistical analysis will be done.

Discussion Results of the study will be discussed compared to other studies.

References

1-Jannati Y, Bagheri-Nesami M, Sohrabi M, Yazdani-Cherati J, Mazdarani S. Factors associated with post-surgical delirium in patients undergoing open heart surgery. Oman Med J. 2014 Sep;29(5):340-5.

ELIGIBILITY:
Inclusion Criteria:Adult patients undergoing open heart surgery. -

Exclusion Criteria: Children, patient refusal.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing open heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2028-10-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-surgical delirium in patients undergoing open heart surgery. | 1 year
  Post-surgical delirium in patients undergoing open heart surgery.

SECONDARY OUTCOMES:
Mortality | 1 year
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hazem I Ahmad Sabry, MB,ChB MD, Principal Investigator — Alexandria University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jannati Y, Bagheri-Nesami M, Sohrabi M, Yazdani-Cherati J, Mazdarani S. Factors associated with post-surgical delirium in patients undergoing open heart surgery. Oman Med J. 2014 Sep;29(5):340-5. doi: 10.5001/omj.2014.91. PMID 25337310